CLINICAL TRIAL: NCT04138173
Title: Enhancing Physical Activity in Patients With Interstitial Lung Disease: an Exploratory Randomized Controlled Trial
Brief Title: Enhancing Physical Activity in Patients With Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S62505
Record Dates: First submitted 2019-10-09; First posted 2019-10-24 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Interstitial Lung Disease; Interstitial Pulmonary Fibrosis
Keywords: physical activity; tele coaching
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele coaching group (Experimental): Coaching with daily interaction with the coaching application, based on an adaptive physical activity goal
  Interventions: Behavioral: Tele coaching intervention
- Usual care group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Tele coaching intervention — A.Education about the importance of PA. During a one-to-one interview with the coach motivation, self-efficacy, barriers, favorite activities and strategies to become more active are discussed.
  B. Step counter providing direct feedback.
  C.A smartphone with a project-tailored application. The application provides automated coaching by displaying an activity goal (number of steps) and feedback on a daily basis. The feedback comes with a graphical presentation. Patients' targets are automatically revised weekly.
  D.Telephone contacts triggered in the case of non-compliance with wearing the step counter, failure to transmit data or failure to progress. Coaches are alerted by a note at the coaches' backend to take contact with the patient if needed.
  Arms: Tele coaching group

SUMMARY:
The level of physical activity (PA) has been shown to be an important predictor for morbidity and mortality in patients with chronic respiratory diseases such as COPD and more recently Idiopathic Pulmonary Fibrosis. Physical inactivity is a common feature of patients with chronic respiratory diseases. Whereas pulmonary rehabilitation is known to result in benefits in exercise capacity, symptoms and quality of life, these gains will not automatically translate into increases in physical activity. Therefore, the present study aims to investigate the effect of a physical activity coaching program on the physical activity level of patients with interstitial lung disease.

DETAILED DESCRIPTION:
The present study aims to

1) primary objective: To explore the magnitude of the effect of a semi-automated tele coaching intervention to enhance physical activity in patients with interstitial lung disease, as measured at 12 weeks, expressed as mean daily step count.

2) Secondary objectives:

1. To test the magnitude of the effect of a 12 weeks coaching intervention on mean time in at least moderate intense activity, walking time, movement intensity, activity bout duration, exercise capacity, quadriceps force and health status.
2. To investigate the patient's experience with this intervention
3. To test the effect of a 12 weeks coaching intervention on the physical activity from a patient experience.
4. To explore the relation between physical activity and vitamin D

Therefore, the study will include stable patients with interstitial lung disease who will be randomized into an intervention (semi-automated coaching intervention) and control (usual care) group. The study consists of a total of 3 visits.

* visit 1: Screening visit
* visit 2: Randomization visits, scheduled 1-2 weeks after visit 1
* visit 3: Follow-up visit, schedules 12 weeks after visit 2

Patients will be randomized into the intervention and control group. In both groups patients will receive information about the importance of being physically active and the physical activity recommendations provided by the world health organization. This information will be provided in a leaflet that will be discussed in an education session (one-to-one) of 10-15 minutes.

1. The control group will receive usual care together with the educational information.
2. Patients in the intervention group will receive a multicomponent tele coaching intervention that consists of 1) education about the importance of physical activity and a one-to-one interview with the coach discussing motivation and barriers to be active, 2) a step counter providing direct feedback, 3) application installed on a smartphone providing an adaptive goal and daily and weekly feedback and 4) contact with the coach if the patient is not compliant with the intervention or not increasing physical activity. The patient is asked to have a daily interaction with the smartphone application.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients, older than 18 year, with a diagnosis of interstitial lung disease
2. Understand and able to work with a smartphone application, as judged by the investigator
3. On stable pharmacotherapy
4. DLCO ≥30%predicted

Exclusion Criteria:

1. On the waiting list for a lung transplantation
2. Life expectancy below 3 months
3. Respiratory tract infection or an exacerbation or change in maintenance medication within 4 weeks before study enrolment
4. Extra pulmonary impairments, unrelated to the underlying lung disease, interfering with physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Daily number of steps at 12 weeks | 12 weeks
  Change in weekly mean step count 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer (Dynaport Movemonitor) validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis. A measurement will be considered valid when having more than four valid days.

SECONDARY OUTCOMES:
Time spent in at least moderate intense activity | 12 weeks
  Change in daily time spent in at least moderate intense activity 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Mean walking time per day | 12 weeks
  Change in mean daily walking time 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Movement intensity | 12 weeks
  Change in mean movement intensity 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Activity bout duration | 12 weeks
  Change in mean duration of an activity bout 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Exercise capacity | 12 weeks
  Change in six-minutes walk distance 12 weeks post randomization in the intervention group as compared to the control group. The six-minute walking test will be performed with standardized encouragement to assess patients' functional exercise capacity. The best of two measurements will be used.
Maximal voluntary isometric quadriceps force | 12 weeks
  Change in isometric quadriceps force 12 weeks post randomization in the intervention group as compared to the control group. The quadriceps isometric strength will be evaluated by a maximal voluntary contraction using the Biodex, a computerized dynamometer. Patients will be seated with a 90° hip and 60° knee flexion. The best of 3 measurements will be taken into analysis as the maximal force capacity of the lower limb.
Health status | 12 weeks
  Health status will be measured by the The King's Brief Interstitial Lung disease (K-BILD) questionnaire. The K-BILD questionnaire is a valid self-completed health status measure for patients with interstitial lung disease consisting of 15 items that measures health status in 3 domains (Psychological, Breathlessness and activity and chest symptoms) and a total score.
Symptoms of anxiety and depression | 12 weeks
  Symptoms of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADs). The HADs is a generic screening measure of symptoms of anxiety and depression. The HADS is a 14 item measure comprising 7 anxiety items and 7 depression items from which separate anxiety and depression sub-scale scores are calculated.

OTHER OUTCOMES:
Physical activity from a patient's perspective (Exploratory endpoint) | 12 weeks
  The c-PPAC, a 12-item questionnaire assessing physical activity from a patient's perspective reflecting the past 7 days will be collected. The questionnaire investigates the amount of and difficulty with physical activity as perceived by the patient. The 2 domain scores (i.e. amount and difficult) as well as the total score will be retrieved as outcomes.
Time to first hospital admission | 2 year
  For explanatory purposes, time to first hospital admissions will be collected in these patients in the 2 years following on the present study.
Transplantation free survival | 2 year
  For explanatory purposes, transplantation free survival status will be collected in these patients in the 2 years following on the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Trooosters, Prof, Principal Investigator — KU Leuven; Heleen Demeyer, Prof, Principal Investigator — KU Leuven; Wim Janssens, Prof, Principal Investigator — KU Leuven; Wim Wuyts, Prof, Principal Investigator — KU Leuven
Locations (1):
- KULeuven, Leuven, Belgium

REFERENCES:
- [Derived] Breuls S, Zlamalova T, Raisova K, Blondeel A, Wuyts M, Dvoracek M, Zurkova M, Yserbyt J, Janssens W, Wuyts W, Troosters T, Demeyer H. Physical activity coaching in patients with interstitial lung diseases: A randomized controlled trial. Chron Respir Dis. 2024 Jan-Dec;21:14799731241235231. doi: 10.1177/14799731241235231. PMID 38511242